CLINICAL TRIAL: NCT06317194
Title: A Novel Method of Non-Invasive Brain Stimulation (Kilohertz Transcranial Magnetic Perturbation) to Enhance Motor Function in Chronic Stroke Patients
Brief Title: A Novel Method of Non-Invasive Brain Stimulation (kTMP) to Enhance Motor Function in Chronic Stroke Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Magnetic Tides (Industry)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Magnetic Tides
Record Dates: First submitted 2024-03-05; First posted 2024-03-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: kTMP; Motor Rehabilitation; Ischemic Stroke; Hemorrhagic Stroke; Cerebrovascular disease; Cortical Excitability; Plasticity; Neuroscience; Stroke; Central Nervous System Disease; kilohertz Transcranial Magnetic Perturbation
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Cerebrovascular Disorders; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active kTMP (Experimental): Participants received 2-8 V/m of active stimulation
  Interventions: Device: kTMP
- Sham kTMP (Sham Comparator): Participants received 0.01 V/m of sham stimulation
  Interventions: Device: Sham kTMP

INTERVENTIONS:
Device: kTMP — A new non-invasive brain stimulation tool
  Arms: Active kTMP
Device: Sham kTMP — A new non-invasive brain stimulation tool with sham setting selected
  Arms: Sham kTMP

SUMMARY:
Stroke is a leading cause of disability with many patients suffering chronic motor function impairments that affect their day-to-day activities. The goal of this proposal is to provide a first assessment of the efficacy of an innovative non-invasive brain stimulation system, kTMP, in the treatment of motor impairment following stroke.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test and validate a novel first-in-class non-invasive approach to enhance motor function in chronic stroke patients. The kilohertz Transcranial Magnetic Perturbation (kTMP) device allows the investigators to target frequency-specific neural activity non-invasively - with no patient discomfort - at and beyond stimulation intensities associated with enhanced recovery from stroke (up to 8 V/m), something that is not possible to achieve with existing NIBS methods.

The trial aims to evaluate the preliminary efficacy of kTMP in improving upper limb motor performance in patients suffering from chronic stroke. This clinical trial aims to target the perilesional motor cortex to assess both immediate and long-term improvement of motor performance, and corresponding physiological changes induced by kTMP stimulation.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 or older with stable upper limb motor dysfunction caused by a single ischemic and/or hemorrhagic stroke greater than 6 months prior to recruitment
2. Fugl-Meyer Assessment: Upper Extremity (FMA UE) score 28-60
3. Motor evoked potentials in a hand muscle when stimulating ipsilesional cortex with suprathreshold single-pulse TMS (MEP+), a proxy of residual corticospinal function.

Exclusion criteria:

1. Participants with cognitive impairment (MoCA < 20), language impairment that interferes with their ability to adhere to the protocol or to provide informed consent.
2. Individuals who are pregnant, have uncontrolled medical problems including but not limited to severe cardiovascular and cardiopulmonary disease, severe alcohol or drug abuse within the past year, or major depression.
3. Contraindications related to non-invasive brain stimulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Fugl- Meyer Assessment (Upper Extremity) | 10 months
  A comprehensive clinical examination that has been widely used to evaluate stroke-related motor impairment. It is graded from 0 (hemiplegia) to 66 for the Upper extremity. Higher scores signifies better motor control, and hence a better outcome.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | 10 months
  A standardized assessment of functional hand motor performance measured by four basic movements used in everyday life (gross arm movement, grasp, grip and pinch). The scores range from 0 to 57. Higher score means a better arm motor status.
Modified Ashworth Scale (MAS) | 10 months
  Used to measure spasticity in wrist and hand flexors and extensors. It assigns a grade of spasticity from 0-4. Lower scores represent normal muscle tone and higher scores represent spasticity. Hence lower scores are associated with better outcomes.
Trial to Trial Variability (T2TV) | 10 months
  Defined as the mean-squared error between the joint angle time-series for a given trial and the median joint angle timeseries. The median T2TV will be calculated for eleven degrees of freedom.
Range of Joint Motion (ROM) | 10 months
  defined as the standard deviation of the joint angle time series for a given trial. The median ROM will be calculated for eleven degrees of freedom and then averaged. If there are joints which appear to be compensatory, they will be removed from the analysis
Grasp to Lift Time | 10 months
  Calculated for each of three epochs, pre, during and post
Transport Time | 10 months
  Calculated for each of three epochs, pre, during and post

CONTACTS AND LOCATIONS:
Locations (1):
- Magnetic Tides, El Cerrito, California, United States

IPD SHARING:
Plan to Share IPD: No